CLINICAL TRIAL: NCT06492811
Title: A Prospective, Randomized, Double-blind Clinical Trial to Evaluate the Efficacy and Safety of a Hydrogel Containing Cascade Catalytic Enzymes in the Treatment of Diabetic Wounds
Brief Title: Efficacy and Safety of a Hydrogel Containing Cascade Catalytic Enzymes in the Treatment of Diabetic Wounds
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of University of South China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: nhfy20240305
Record Dates: First submitted 2024-07-01; First posted 2024-07-09 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Diabetic Wound

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- GAT@F nanoenzyme hydrogel complex (Experimental): The glucose oxidase (GOx) and catalase (CAT) cascade systems have been included in the therapeutic system of diabetic wounds,with GOx primarily consumes glucose to create H2O2, while CAT further catalyzes H2O2 to provide sufficient oxygen.Natural enzymes have excellent cascade catalytic efficiency as well as biocompatibility. Hydrogels have high water content and cargo loading efficiency, as well as superior biocompatibility, making them popular in wound healing applications.
  Interventions: Drug: GAT@F nanoenzyme hydrogel complex
- Medical chitosan bio-gel dressing (Active Comparator): The medical device database of the National Medical Products Administration (NMPA) was searched and the Medical chitosan bio-gel dressing (6S YinYu)(20182640080) was selected.
  The positive control product used in this trial is based on the following points:
  1. The properties of the test products are similar, and both the test products and the control products are hydrogel dosage forms;
  2. In terms of the duration of therapeutic effect, both the experimental product and the control product could achieve the maintenance of therapeutic effect;
  3. The control product is widely used by clinicians at this stage, and its clinical efficacy is relatively confirmed, with good clinical effect and safety, and it is one of the treatment products recognized by the industry for wound repair.
  Interventions: Drug: GAT@F nanoenzyme hydrogel complex
- Blank hydrogel dressing (Placebo Comparator): Hydrogel dressings can maintain a moist environment at the wound site, which promotes cell migration and tissue regeneration, thus accelerating the healing process. Hydrogels have excellent absorption capabilities, helping to manage wound exudate and reduce the risk of infection by forming a physical barrier against bacteria and contaminants. Moreover, hydrogels are biocompatible and unlikely to cause allergic reactions or rejection. Their softness and flexibility enable them to conform to irregular wound surfaces, providing effective coverage and protection.
  Interventions: Drug: GAT@F nanoenzyme hydrogel complex

INTERVENTIONS:
Drug: GAT@F nanoenzyme hydrogel complex — The wound condition was recorded by taking photos each time the dressing was changed. The diabetic wound was routinely treated with a dressing change, after which GAT@F nanoenzyme hydrogel complex was applied externally and a secondary dressing - medical surgical gauze was added. According to existing clinical data, it is recommended to use no more than 10ml per dressing change.

SUMMARY:
This clinical study is a prospective, randomized, double-blind, positive-controlled, parallel study. Subjects who sign study informed consent (ICF) approved by Ethics Committee (EC) and meet all of the inclusion criteria and none of the exclusion criteria are eligible to enter the study.This clinical study is expected to include 49 participants and treat patients with diabetic wounds.Each participant is expected to participate for about 3 months, including a 2-week screening period, a 2-week dressing period, and an 8-week safety follow-up period.

Successfully enrolled subjects will be randomly divided into one of the following treatment groups: (1)GAT@F nanoenzyme hydrogel complex dressing(2)Medical chitosan bio-gel dressing (3)Blank hydrogel dressing.

Diabetic wounds were treated with experimental dressing, and dressing was changed once a day for 14 consecutive days.Neither subjects nor investigators were informed of the treatment assignment.During treatment, the granulation coverage rate and wound healing rate of each group were evaluated at the second visit, the third visit and the fourth visit.Wounds were scored using Wagner grading scale, Wlfl grading scale and IDSA/IWGDF grading scale.The histological morphology, ROS, sugar content, IL-6 and TNF-α of the wound were quantitatively detected at the second and fifth visits, and the changes of the data results compared with baseline were evaluated.The tolerability (occurrence of local adverse events) and acceptability (ease of application and removal, adherence of the dressing to the wound bed, bleeding or pain during dressing removal) of the dressing were qualitatively assessed and recorded at the 2nd visit, 3rd visit, and 4th visit.The safety follow-up was conducted by telephone on the 30th and 60th day after the last treatment to collect safety information.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who voluntarily participate in this clinical study and sign informed consent;
2. Subjects aged 18-80 years (including boundary values), male or female;
3. Participants must meet the following criteria to participate in the study:

   1. Female subjects:

      * Nonfertile (biologically incapable of becoming pregnant, including women who have gone through menopause for more than 2 years)
      * Be potentially fertile, have a negative pregnancy test result, and agree to adhere to the correct use of an acceptable and effective contraceptive method during the study period
   2. Male subjects:

      * An effective form of contraception or an effective form of contraception by a partner of the opposite sex must be used during the period of participation in this clinical trial 4)The clinical manifestations of the patient can meet the diagnostic criteria of diabetes; 5)There was at least 1 month of unhealed wounds before joining the clinical trial; 6)The patient's blood glucose was controlled at fasting blood glucose < 8mmol/L and at 2 hours after meal blood glucose < 11.1mmol/L; 7)Diabetic wounds meet Wagner grades 1 to 2; 8)Diabetic wounds conform to IDSA/IWGDF grade ≤2; 9)Diabetic wounds conform to the Wlfl evaluation system rating ≤2; 10)The size of the wound area is between 9cm2 and 100cm2; 11)There was a history of surgical dressing change or a desire for surgical intervention within 1 month before the visit; 12)In the investigators' judgment, subjects were willing and able to adjust the current diabetic wound treatment regimen as required; 13)Subjects must be willing to complete all visit assessments as required by the study protocol.

Exclusion Criteria:

Participants in this clinical trial will not be enrolled if they meet any of the following criteria:

1. The subject had any condition that required treatment or that the investigator felt might interfere with the study parameters, including aortitis, deep vein thrombosis, arterial thromboembolism, thromboangiitis obliterans, and varicose veins of the lower extremity; Patients with spinal cord injury and syringomyelia;
2. Patients who have been diagnosed with chronic wounds caused by autoimmune diseases such as Becset's disease, psoriasis, or pemphigus, or who have used immunosuppressive biologics or immunosuppressants within the last 12 months or are expected to use them during the study period;
3. Any lower extremity vascular and related surgery is planned during the study period;
4. Women who are pregnant or breastfeeding or plan to become pregnant during the study period, or women who are fertile but not using effective contraception;
5. Patients with pacemakers, severe weakness of heart, lung and kidney function, malignant tumors, various bleeding disorders, acute infectious diseases, high fever, high fever disease, cardiac surgery after recovery, or have a medical condition that the physician believes may prevent the subject from participating in the study and follow-up;
6. The subject is allergic to the same dressing;
7. Subjects had a history of alcohol and drug abuse;
8. Subjects have significant medical conditions other than diabetic wounds (sepsis, tuberculosis, etc.), trauma, or other conditions that, in the investigator's judgment, would put them at risk for participating in the study, or would interfere with the study results, or would have an illness or condition that would affect their ability to participate in the study;
9. Antibiotic dressings, silver ion dressings, zinc ion dressings and other dressings that interfered with the study results were used within 14 days prior to enrollment;
10. The investigator, the assisting investigator, the investigator participating in the study, and the immediate family of the person mentioned above;
11. History of mental illness, mental retardation, or other medical conditions that affect the validity of informed consent in this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Granulation coverage | 14 days
  Wound granulation tissue coverage (%) = (granulation coverage area)/(total wound area) ×100%

SECONDARY OUTCOMES:
Wound healing rate | 14 days
  Wound healing rate (%) = (original wound area - current wound area)/(original wound area) ×100%
Wagner rating Scale | 14 days
Wlfl rating Scale | 14 days
IDSA/IWGDF rating scale score | 14 days
Histopathological analysis score | 14 days
ROS quantitative detection value of wound tissue | 14 days
Quantitative measurement of sugar content in wound tissue | 14 days
Quantitative detection of IL-6 and TNF-α in wound tissue | 14 days

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of University of South China, Hengyang, Hunan, China

IPD SHARING:
Plan to Share IPD: No